CLINICAL TRIAL: NCT05523349
Title: An Investigation on Function and Performance of a New Microprocessor-controlled Prosthetic Knee
Brief Title: An Investigation on Function and Performance of a New Microprocessor Controlled Prosthetic Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Össur Iceland ehf (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP2022022514
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Prosthesis User; Amputation

STUDY DESIGN:
Intervention Model Description: Considering previous experience with clinical investigations in prosthetics it was concluded to conduct a non-randomized prospective repeated measures (ABA) design, comparing subjects' current MPK at baseline and 3-week follow-up vs. the investigational device at 3-week follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- NAVii (Experimental): Users will be fitted with a new microprocessor-controlled prosthetic knee for 3 weeks to compare to their usual device.
  Interventions: Device: NAVii

INTERVENTIONS:
Device: NAVii — Passive Microprocessor-controlled prosthetic knee

SUMMARY:
This investigation aims to compare the functional performance of a new passive microprocessor-controlled Prosthetic Knee to subjects usual microprocessor-controlled prosthetic knee.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of the investigational device compared to other passive MPKs (Rheo Knee 4, C-leg 4, Genium, X3, Plié 3, Orion 3, Quattro, Allux) regarding satisfaction in descending activities for moderate to high active prosthesis users within the intended population for the investigational device.

Additionally, to evaluate the balance confidence, perception of safety and comfort in standing with the investigational device compared to other passive MPKs (Rheo Knee 4, C-leg 4, Genium, X3, Plié 3, Orion 3, Quattro, Allux).

In phase I the performance in descending activities will be compared to any other passive MPK and in phase II there will be a subgroup analysis comparing to hydraulic MPKs and Rheo Knee 3, specifically.

The test will be a non-randomized single group open label prospective repeated measures (ABA) design.

Amputees are a small proportion of the general population. The population group specified in the inclusion/exclusion criteria is a further subsample of amputees. For practical reasons, i.e. to achieve statistical power, it is therefore more feasible to use within-subject comparison rather than creating study arms to compare. Furthermore, as mobile amputees generally have and use a prosthetic device for their daily activities, within-comparison is feasible comparing to the subject's previous device.

All investigational activities will be conducted at prosthetic out-patient clinics.

As stated above the primary endpoint is Satisfaction on descending stairs, and the secondary endpoints are satisfaction on descending ramps, balance confidence and standing comfort in that respective order of significance. In addition, there are two exploratory endpoints on mobility and balance during ambulation.

Procedures:

i) Recruitment Potential subjects will be identified from the customer base of the Local Principal Investigator (LPI). LPI evaluates, based on previous experience of interaction with and servicing of patients, if a potential participant is cognitively capable. If a potential participant fits the inclusion and exclusion criteria the LPI will contact them via telephone. During the telephone call the LPI will verify if they are interested in participating in a study. If interest is expressed at this point they will answer some screening questions and if the eligibility criteria are met an appointment will be made for the clinical visit and signing of the ICF. Questions relating to the duration of the study, number of clinical visits required and the investigational device will be answered.

Potential risk of participating in the investigation will be explained to the subject at this point to the candidate for enrolment.

The LPI will communicate to the study monitor and sponsor co-investigator the number of users he has identified that meet the inclusion criteria and are willing to participate.

ii) Test procedure There are three scheduled study events. Three sites will be included in the study, 4-10 users will be recruited at each site. At the initial visit, the first study event, for each subject a researcher qualified to obtain informed consent will seat the subject and proceed as described.

Prior to fitting the subject will be asked to provide feedback on the current prosthesis, by filling in a set of questionnaires (Including background information) and perform functional tests. The users will be fitted within the standard methods of prosthetic fitting, alignment, introduction, training and walking on various terrain.

After initial fitting, subjects will receive standard training on the investigational device by a certified prosthetist (the LPI) with support from sponsor investigators. When training is complete, and subjects feel comfortable and safe they will leave the site on the investigational device to use as their primary prosthesis in their daily life for 3 weeks. During this 3 week period the LPI will be in weekly contact with subjects via telephone to check on any issues that may arise.

The second visit will be at three weeks after visit 1. During this visit subjects will complete the same functional tests and questionnaires as at visit 1 (excluding background information) on the investigational device, with the addition of a usability questionnaire. They will then be fitted back to their prescribed device.

The third visit will be three weeks later. During this visit subjects will complete the same functional tests and questionnaires as at visit 2 (excluding usability questionnaire) on their prescribed device, as well as completing a qualitative interview on their experiences with both microprocessor knee devices.

iii) Measurements and data collection The same questionnaires, consisting of three valid instruments (PEQ questions, PLUS-M and ABC), will be used and filled in at three separate points in time. Background information will be collected at baseline only, usability questionnaire at visit 2 only and qualitative interview at visit 3 only. An activity report will be generated from the investigational device at visit 2 and an activity report from subjects prescribed device at visit 3, if applicable.

ELIGIBILITY:
Inclusion Criteria:

* 45Kg< body weight < 136Kg
* Cognitive ability to understand all instructions and questionnaires in the study;
* Unilateral TF/KD amputees that are regular prosthesis users for at least 3 months
* Current MPK users (passive MPKs only)
* Age ≥ 18 years
* Willing and able to participate in the study and follow the protocol
* Moderate to high active users (PLUS M T-score>4021)

Exclusion Criteria:

* Users with stump pain
* Users with socket problems
* Pregnant Users
* Users using Power Knee, Kenevo or mechanical knees as their prescribed prosthesis
* Alignment that cannot be matched with the Rheo Knee 4 setup, as described in Instructions for use.
* Osseointegration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt N Gruben, CPO, Principal Investigator — Ossur Americas
Locations (4):
- United States (3):
  - Bionic P & O, Merrillville, Indiana
  - Oakland Orthopedic appliances, Bay City, Michigan
  - Perry Prosthetics, Perrysburg, Ohio
- Ossur Motionlab, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Users will be fitted with a new microprocessor-controlled prosthetic knee for 3 weeks to compare to their usual device.
  NAVii: Passive Microprocessor-controlled prosthetic knee
Period: Overall Study
Arm/Group | All Participants
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
  Iceland | 2
PLUS-M T-Score [Mean (Standard Deviation); unit: T-score] — Prosthetic Limb Users Survey of Mobility (PLUS-M), self-report instrument measuring mobility of adults with lower limb amputation. Scoring a PLUS-M short form produces a T-score. T-score equals the sum for all responses on the short form (creating a raw score). raw score needs to be used to determine the T-score in the conversation table provided with the PLUS-M questionnaire. The T-score is a standardized score with a mean of 50 and a standard deviation of 10. A higher T-score indicates a higher level of mobility. The highest possible T-score is 71.4 and the lowest one is 21.8.
  T-score | 55.3 (4.9)
Socket Comfort Score [Mean (Standard Deviation); unit: scores on a scale] — self-report; the amputee rates their socket comfort on a 10-point Likert scale where 0 is "most uncomfortable" and 10 is "most comfortable". It is assumed that for subjects with a score of 5 or lower the socket comfort is too low and may affect other study parameters.
  scores on a scale | 9.1 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction During Stair Descent
Description: A question from the Prosthesis Evaluation Questionnaire (PEQ) regarding the satisfaction of walking downstairs is answered; scale allows for values from 1 to 10 while 1 represents very low satisfaction and 10 high satisfaction. The analysis was done by using a Bayesian approach which presents the posterior distribution of effects between Visit 2 and visit 3. The parameter for analysis is the difference of the score between Visits 2 and 3. If scores in Visit 2 (subjects using the investigational device) were larger than in visit 3 (subjects using their prescribed device), the difference of Visit3 - Visit2 scores would be negative and would therefore support the corresponding hypotheses. The Median difference and range of the Confidence interval of the difference are reported in the outcome measure data table.
Time Frame: for analysis data from visit 2 (3 weeks after visit 1) and visit 3 (3 weeks after visit 2) were used
Measure: Median (89% Confidence Interval); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 14
score on a scale | 0.80 [-0.50 to 2.1]

2. Secondary Outcome: Six Minute Walk Test
Description: The Six Minute Walk test (6MWT) is a record of the distance traveled by a given patient at his or her self-selected walking speed over a period of six minutes. All that is required is a stopwatch and a walking corridor or track of known distance.
Time Frame: for the final analysis data from visit 2 (3 weeks after visit 1) and visit 3 (3 weeks after visit 2) were used
Population: One subject had only limited lung function. At the first visit, the subject wanted to give it a try to walk the full 6 minutes, but the measurement was aborted by the investigators as the test was considered too demanding. The 6 MWT was skipped for that subject in the consecutive visits.
  One subject did not complete the 6 MWT at the last visit with Rheo knee as the subject reported on functional issues of the knee. Their CPO has taken care of the issue.
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | All Participants
Number analyzed (Participants) | 12
meter
  Visit 2 | 326.8 (90.7)
  Visit 3 | 326.7 (82.6)

ADVERSE EVENTS:
Time Frame: adverse event data were collected over the time of participation starting with the first visit until the third visit (6 weeks for each participant)
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=14)
Fall (Social circumstances) | 1 (1) — subject fell after a friend had switched off the device as a joke

LIMITATIONS AND CAVEATS:
Prosthetic use time was not monitored or controlled for during the adaptation time period, the actual time each subject used the investigational device is therefore unknown.

The sample of the trial represents only a small portion of the whole population with above knee amputation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT05523349/Prot_SAP_000.pdf